CLINICAL TRIAL: NCT02468050
Title: Effectiveness of Exercise Training and Self Management in the Attenuation of Anxiety and Depressive Symptoms Following Breast Biopsy
Brief Title: Study of Exercise to Manage Distress During Breast Screening
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 17796
Record Dates: First submitted 2012-06-25; First posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer; Anxiety; Depression
Keywords: Anxiety; Depression; Exercise; Breast Cancer; Biopsy; Screening; Diagnosis
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders; Depression; Motor Activity; Disease | interventions — Exercise; Self-Management; Professional Autonomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Self Management (Experimental): In addition to the weekly supervised exercise session, participants in this arm will view an instructional video. The video will deliver theory driven training of cognitive behavioural strategies for self management of exercise. It is expected that this will improve adherence to the exercise program.
  Interventions: Behavioral: Moderate intensity exercise training; Behavioral: Self Management of exercise
- Exercise (Experimental): Personalized 6 week moderate intensity (50 - 75% of heart rate reserve) facility and home based exercise program including cardiovascular and muscular conditioning.
  Interventions: Behavioral: Moderate intensity exercise training
- Prospective Cohort Control (No Intervention): Eligible, consented participants who are unable to attend the weekly exercise sessions will serve as a cohort control group. Participants will be asked to complete patient reported measures of anxiety, depression, and exercise behaviour within 3 days of biopsy, and 6 weeks post biopsy.

INTERVENTIONS:
Behavioral: Moderate intensity exercise training — 6 weeks of moderate intensity exercise training (50 - 75% of heart rate reserve). Sessions are facility and home based and include cardiovascular warm-up, cardiovascular training, muscular conditioning, and flexibility exercises.
  Other Names: Exercise; Treatment Group 1
  Arms: Exercise; Self Management
Behavioral: Self Management of exercise — In addition to the 6 week exercise program (refer to Exercise Treatment Group), participants randomly assigned to the Self Management Group will learn strategies for the self management of exercise.
  Other Names: Self Management; Self Regulation; Adherence; Treatment Group 2
  Arms: Self Management

SUMMARY:
The breast cancer screening and diagnostic period is associated with heightened symptoms of anxiety and depression. Physical exercise has been found to effectively decrease these symptoms in healthy and diseased populations. This study aims to determine if a pre treatment exercise intervention can minimize symptoms of anxiety and depression in women undergoing screening for breast cancer.

DETAILED DESCRIPTION:
The breast cancer diagnostic process is associated with anxiety and depression. Physical exercise has emerged as an attractive non-pharmacologic approach to mitigating the psychological and physical sequelae of breast cancer and its treatments, however pre treatment interventions are not integrated into current practice. This study aims to determine the effectiveness and feasibility of a pre treatment exercise intervention in attenuating levels of anxiety and depression following breast biopsy and throughout the diagnostic period.

ELIGIBILITY:
Inclusion Criteria:

* undergoing breast biopsy at St. Joseph's Health Care, London Ontario
* minimum BI-RADS 4a
* physically inactive

Exclusion Criteria:

* meeting Health Canada Guidelines for Physical Activity for past 6 months
* medical contraindications to exercise
* unable to participate in moderate intensity exercise program

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Symptoms of anxiety will be assessed using patient reported anxiety inventory | Change in baseline (within 1 week of breast biopsy) at Week 3 and at Week 6
  Spielberger State-Trait Anxiety Inventory - State Form (STAI; Spielberger, Gorsuch, & Lushene, 1970).

SECONDARY OUTCOMES:
Symptoms of subclinical depression will be assessed using a patient reported inventory | Within 1 week of breast biopsy, Week 3, Week 6
  Centre for Epidemiologic Studies-Depression Scale (CES-D; Radloff, 1977).
Exercise behaviour will be assessed using a patient reported inventory | Within 1 week of breast biopsy, Week 3, Week 6
  Leisure Time Exercise Questionnaire (Godin & Shephard, 1985)
Body composition: Dual X-Ray Absorptiometry scan (GE Lunar iDXA) | Baseline (within 1 week of breast biopsy), Week 6
Self Efficacy: patient reported inventory assessing efficacy for self management of exercise | 1 week post breast biopsy, Week 3, Week 6
Optimism: patient reported inventory assessing dispositional optimism | Baseline (within 1 week of core breast biopsy)
  Life Orientation Test-Revised (LOT-R; Scheier, Carver, & Bridges, 1994).
Symptoms of dispositional anxiety will be assessed using patient reported anxiety inventory | Within 1 week of breast biopsy
  STAI - Trait Form

CONTACTS AND LOCATIONS:
Overall Officials: Muriel Brackstone, MD PhD FRCSC, Study Director — London Regional Cancer Program; Anita G Cramp, PhD, Study Director — Western University; Amy Kossert, MHK, Study Director — Western University; Harry Prapavessis, PhD, Principal Investigator — Western University
Locations (1):
- Exercise and Health Psychology Laboratory, Western University, London, Ontario, Canada